CLINICAL TRIAL: NCT02039609
Title: Nutritional Metabolomics: the Search for Dietary Exposure Variables 2
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Nutritional Metabolomics AIKN2
Record Dates: First submitted 2013-12-17; First posted 2014-01-17 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: vegetarian; vegan; omnivore; Habitual diet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Omnivores: No intervention, habitual diet
- Vegetarians: No intervention, habitual diet
- Vegans: No intervention, habitual diet
- Vegetarians consuming fish: No intervention, habitual diet

SUMMARY:
In the post-genomic era, a major challenge for health research is to understand the complex interactions among genetic, environmental and lifestyle factors including dietary intake. Unfortunately, such initiatives are hampered by the lack of accurate dietary intake assessment methods for large studies. The newly emerging field of metabolomics offers unique possibilities to characterize individual food intake, dietary patterns and effects of dietary intervention in large studies. The investigators propose to develop a platform to detect broad metabolomic responses to food intake in controlled trials as well as to use targeted metabolomics approaches to characterize dietary intake in longitudinal studies. Our laboratory has a long history of developing methodology for assessing nutritional status and effects of diet on metabolism. Here, the investigators team up with the Sahlgrenska Academy Core Facility and the Swedish NMR Centre at the University of Gothenburg, that offer modern metabolomics equipment and competence in bioinformatics, and use this in the context of nutrition research. To their knowledge, the investigators are among the first groups in the country to develop skills in metabolomics to assess dietary intake and effects of nutrition on metabolism, and probably the first to use two complementary platforms with both mass-spectrometry and nuclear magnetic spectroscopy. Hence, our methodological results should be useful to nutritional scientists nationally as well as internationally.

ELIGIBILITY:
Inclusion Criteria:

Healthy Body mass index 18.0-30.0, age 18-65 yrs

Exclusion Criteria:

Regular Medication or tobacco use Pregnancy or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects Adults
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Metabolomic patterns that reflect habitual diet | Fasting blood sample in the morning at one occasion
  Long-time vegans, vegetarians and omnivores will be asked to donate a fasting blood sample at one occasion, in the early morning. This blood sample will be analyzed, using nuclear magnetic resonance (NMR) and mass spectrometry (MS) techniques to reveal all metabolites. Patterns among these metabolites will be distinguished using the statistical techniques principal component analysis and discriminant analysis.

SECONDARY OUTCOMES:
Discriminating vegan-, vegetarian- and omnivorous diets by hair isotopic analysis | Hair samples in the morning at one occasion
  The same study group also was asked to donate 5-10 hairs of 2 cm closest to the scalp. These were analyzed using isotope ratios of 15N and 13C by IRMS, to see if also this method could discriminate between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Anna K Winkvist, PhD, Principal Investigator — Univ of Gothenburg, Sweden; Lars H Ellegard, PhD, MD, Study Chair — Univ of Gothenburg, Sweden; Helen M Lindqvist, Study Director — Univ of Gothenburg, Sweden
Locations (1):
- Dept Internal Medicine and Clinical Nutrition, Univ of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Lindqvist HM, Radjursoga M, Torstensson T, Jansson L, Ellegard L, Winkvist A. Urine Metabolite Profiles and Nutrient Intake Based on 4-Day Weighed Food Diary in Habitual Vegans, Vegetarians, and Omnivores. J Nutr. 2021 Jan 4;151(1):30-39. doi: 10.1093/jn/nxaa019. PMID 32047921
- [Derived] Lindqvist HM, Radjursoga M, Malmodin D, Winkvist A, Ellegard L. Serum metabolite profiles of habitual diet: evaluation by 1H-nuclear magnetic resonance analysis. Am J Clin Nutr. 2019 Jul 1;110(1):53-62. doi: 10.1093/ajcn/nqz032. PMID 31127814